CLINICAL TRIAL: NCT04069975
Title: Sedation Versus No Sedation for Diagnostic Esophagogastroduodenoscopies and Detection Rates of Precancerous Lesions and Cancer: a Case-control Study
Brief Title: Sedation Versus No Sedation for Detection Rates of Precancerous Lesions and Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Collaborators: Weihai Municipal Hospital (Other); Binzhou Medical University (Other); Qilu Hospital of Shandong University (Qingdao) (Other)
Responsible Party: Principal Investigator, Yanqing Li, Professor, Shandong University
Other Study IDs: 2019SDU-QILU-09
Record Dates: First submitted 2019-08-24; First posted 2019-08-28 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Early Detection of Cancer
Keywords: Early Detection of cancer; Gastrointestinal Neoplasms; Endoscopy, Gastrointestinal
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No sedation: The group of patients who did endoscopies without sedation.
- Sedation: The group of patients who did endoscopies with sedation.
  Interventions: Other: Sedation

INTERVENTIONS:
Other: Sedation — The group of patients who did endoscopies with or without sedation. (This is a choice of themselves)
  Groups: Sedation

SUMMARY:
The influence of sedation on the endoscopic detection rate of the precancerous lesions and cancer of upper digestive system has not been assessed. In the daily medical routine of China, patients have the right to choose the sedation style according to his or her own situation, whose detailed endoscopic data of patients are recorded in the endoscopy quality control system. The aim of this research is to detect whether the use of sedation can help improve detection rate of precancerous lesions and cancer of upper digestive system.

DETAILED DESCRIPTION:
The influence of sedation on the endoscopic detection rate of the precancerous lesions and cancer of upper digestive system has not been assessed. In the daily medical routine of China, patients have the right to choose the sedation style according to his or her own situation, whose detailed endoscopic data of patients are recorded in the endoscopy quality control system. The aim of this research is to detect whether the use of sedation can help improve detection rate of precancerous lesions and cancer of upper digestive system.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged more than 18 years with or without GI symptoms attending for endoscopy from 2012 to 2019.

Exclusion Criteria:

* Patients unable to cooperated the endoscopy or unable to complete it. People with endoscopy contraindications are naturally excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: After calulating, the sample size should be more than the largest number 23,000.
  As a retrospective study, the sample size may be more than 20,0000, according to our estimates.
Sampling Method: Probability Sample
Enrollment: 200000 (Estimated)
Dates: Start 2019-06-02 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Detection rate of precancerous lesions and cancer of upper digestive system improvement | 2020
  Detection rate of precancerous lesions and cancer of upper digestive system improvement

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China

REFERENCES:
- [Derived] Zhou J, Li Z, Ji R, Wang P, Zhang A, Wu K, Liu C, Niu Q, Chu Y, Su X, Zuo X, Li Y. Influence of Sedation on the Detection Rate of Early Cancer and Precancerous Lesions During Diagnostic Upper Gastrointestinal Endoscopies: A Multicenter Retrospective Study. Am J Gastroenterol. 2021 Jun 1;116(6):1230-1237. doi: 10.14309/ajg.0000000000001201. PMID 34074827